CLINICAL TRIAL: NCT03993496
Title: Intraoperative Assessment of Pulsatile Aneurysm Wall Motion During Endovascular Aneurysm Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Mark Rockley, Co-Investigator, University of Ottawa
Other Study IDs: 20190366-01H
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Aortic Aneurysm; Endovascular Abdominal Aortic Aneurysm Repair; Ultrasound
Keywords: Abdominal Aortic Aneurysm; Endovascular Abdominal Aortic Aneurysm Repair; Ultrasound; M-mode; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EVAR Patients: Patients with infrarenal abdominal aortic aneurysm scheduled for elective endovascular aneurysm repair (EVAR) surgery will undergo intraoperative assessments of aneurysm wall pulsatility using ultrasound M-Mode.
  Interventions: Diagnostic Test: Abdominal Aortic Aneurysm Sac Pulsatility

INTERVENTIONS:
Diagnostic Test: Abdominal Aortic Aneurysm Sac Pulsatility — Measurements of aortic wall pulsatility will be performed using trans-abdominal ultrasound through the non-sterile field of the upper abdomen, while the surgeons operate through the groins. The pulsatilty of the aneurysm will then be measured using transverse views in 'M-Mode' of the ultrasound, and measures the aneurysm wall displacement during a cardiac cycle; the minimum diameter (diastole) and maximum diameter (systole) will be measured. These measurements will occur during surgery:
  1. Prior to EVAR deployment
  2. After EVAR deployment, but before balloon affixation to the aortic wall
  3. After EVAR deployment and after affixation
  Other Names: M-Mode Ultrasound

SUMMARY:
Endovascular abdominal aortic aneurysm repair (EVAR) aims to reduce the risk of aneurysm (AAA) rupture by reducing the blood pressure transmitted to the wall of the aneurysm. Aneurysms that remain pressurized despite EVAR may continue to grow, therefore requiring additional surgical interventions. The purpose of this study is to infer the reduction of pressure transmitted to the aneurysm wall by using intraoperative ultrasound ('M-Mode') to assess the pulsatility of the aneurysm wall. The hypothesis is that intraoperative reduction in aneurysm wall pulsatility after EVAR will correlate with improved aneurysm sac size reduction.

DETAILED DESCRIPTION:
Endovascular abdominal aortic aneurysm repair (EVAR) aims to reduce the risk of aneurysm (AAA) rupture by reducing the blood pressure transmitted to the wall of the aneurysm. Unfortunately, this procedure is not always successful, and patients need to return to the operating room for further procedures because the aneurysm wall remains pressurized and the aneurysm continues to grow. Currently, there is no standard non-invasive way of measuring aneurysm pressure. The purpose of this study is to infer the reduction of pressure transmitted to the aneurysm wall by using intraoperative ultrasound ('M-Mode') to assess the pulsatility of the aneurysm wall. The hypothesis is that intraoperative reduction in aneurysm wall pulsatility after EVAR will correlate with improved aneurysm sac size reduction. This is clinically relevant because physiologic intraoperative feedback of aneurysm pressure may potentially influence surgical decision making in the future, reducing unnecessary re-interventions. This will also improve our understanding of the intraoperative physiologic response to EVAR.

Our primary research question is in patients receiving elective endovascular repair of abdominal aortic aneurysms (EVAR), does the change in intraoperative ultrasound estimated aneurysm wall pressure during EVAR correlate with aneurysm sac size reduction 1 year after surgery? Secondary objectives are to assess correlation between intraoperative ultrasound estimated aneurysm wall pressure and endovascular leaks and aneurysm-related re-interventions.

A prospective, observational, assessor-blinded and surgeon-blinded study will be conducted at the TOH Civic Campus in Ottawa, ON in order to satisfy the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Elective endovascular aneurysm repair (EVAR) surgery
* Infrarenal abdominal aortic aneurysm
* Age greater than 18 years old

Exclusion Criteria:

* Prior abdominal aortic aneurysm procedures
* Inability to visualize aneurysm on ultrasound
* Inability to provide consent
* Irregular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of anyone over the age of 18 years old with an abdominal aortic aneurysm scheduled for elective endovascular abdominal aortic aneurysm repair (EVAR) through the Division of Vascular & Endovascular Surgery at The Ottawa Hospital, Civic Campus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2019-12-09 (Estimated); Study Completion 2020-12-09 (Estimated)

PRIMARY OUTCOMES:
Fractional aneurysm sac size reduction 1 year after surgery | 1 year
  Aneurysm sac size reduction will be measured using surveillance ultrasound 1 year after surgery. Post-operative imaging reports will be accessed through the hospital electronic health records system (EPIC).

SECONDARY OUTCOMES:
Fractional aneurysm sac size reduction 30 days after surgery | 30 days
  Aneurysm sac size reduction will be measured using CTA 30 days after surgery. Post-operative imaging reports will be accessed through the hospital electronic health records system (EPIC).
Endovascular leaks (Type 1, 2, 3, 4) | 30 days
  The presence of endovascular leaks (type 1, 2, 3, 4) will be assessed intraoperatively with a completion angiogram and CTA at 30 days postoperative. Postoperative imaging reports will be accessed through the hospital electronic heath records system (EPIC).
Aneurysm-related re-interventions | 1 year
  Any aneurysm-related complications requiring re-interventions will be noted. If an additional intervention is performed in the same operation, additional measurements of aortic wall pulsatility following intervention will be included. Other post-operative re-interventions will be reviewed through EPIC.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital - Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No